CLINICAL TRIAL: NCT05120661
Title: Elucidating the Role of Human Small Intestine Microbiota in Interpersonal Differences in GLYcemic Responses Upon Consumption of Food Products: A Proof of Principle Study
Brief Title: Elucidating the Role of Human Small Intestine Microbiota in Explaining Differences in Postprandial Glucose Responses
Acronym: GLYSIMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Guido Hooiveld, Principal Investigator, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NL78737.091.21
Record Dates: First submitted 2021-10-11; First posted 2021-11-15 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Metabolic Syndrome; Obesity; Overweight; Microbiota; Small Intestine; Digestion
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Overweight | interventions — Food

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate-rich food product (to be determined) (Experimental): This is a nutritional product, such as bread or cake, containing 50 gram carbohydrates.
  Interventions: Other: food product
- Another carbohydrate-rich food product (to be determined) (Experimental): This is a nutritional product, such as bread or cake, containing 50 gram carbohydrates.
  Interventions: Other: food product

INTERVENTIONS:
Other: food product — a food product containing 50 gram carbohydrates

SUMMARY:
It has been shown that person-specific factors, such as the fecal microbiome, influenced postprandial glycemia. The small intestine is the site of nutrient digestion and absorption. The small intestine microbiota is amendable by dietary changes, and plays a key role in host adaptability to dietary variations. The role of the human small intestine microbiota in regulating postprandial glycemic responses towards food products will be investigated. First a screening will take place with to choose the test products that elicit most differential glucose responses and to select subjects with differential postprandial response to the same food product. The study will be a 6-day randomized cross-over trial with two test days. Four test (food) products, each containing 50 gram carbohydrates, and an oral glucose tolerance test will be provided to participants. Twenty men or women (BMI≥25 kg/m2, 40-75 years old) will be included. The main study parameters/endpoints are the food product-induced plasma glucose responses (iAUC) and the small intestine microbiota.

DETAILED DESCRIPTION:
Rationale: It has been shown that person-specific factors, such as the fecal microbiome, influenced postprandial glycemia. The small intestine is the site of nutrient digestion and absorption. The small intestine microbiota is amendable by dietary changes, and plays a key role in host adaptability to dietary variations. Differences in small intestine microbiota are hypothesized to be key in explaining the interpersonal differences in glycemic responses.

Objective: To investigate the role of the human small intestine microbiota in regulating postprandial glycemic responses towards food products.

Study design: The subjects will wear a continuous glucose monitor during the screening and the study. First a screening (14 days in total) will take place with to choose the test products (2 out of 4) that elicit most differential glucose responses and to select subjects with differential postprandial response to the same food product. Also an OGTT will be performed. The study will be a randomized cross-over trial with two test days (length of trial is 6 days in total). During the trial, the subjects will be intubated with a naso-jejunum catheter.

Study population: Twenty men or women (BMI≥25 kg/m2, 40-75 years old). Intervention (if applicable): Four test (food) products, each containing 50 gram carbohydrates, and an oral glucose tolerance test.

Main study parameters/endpoints: test (food) product-induced plasma glucose responses (iAUC), small intestine microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* BMI≥25 kg/m2
* Age 40-75 years
* Signed informed consent

Exclusion Criteria:

* Having a history of medical or surgical events that may either put the subject at risk because of participation in the study, or influence the results of the study, including diabetes type 1, a swallowing disorder, gastrointestinal or liver disease, renal failure, cancer, nose/throat diseases, gastric bypass surgery, use of anticoagulants;
* Having a bleeding/coagulation disorder, including hemophilia, Von Willebrand disease, Bernard-Soulier, Glanzmann thrombasthenia or thrombocytopenia;
* Use of antibiotics within 2 months of starting the study or planned during the study;
* Use of medication that could influence the study results, such as diabetes treatment;
* Use of pro- and prebiotic supplements;
* Sensitive to medical skin adhesives;
* Having an allergy or intolerance towards compounds in the test products;
* Follows a vegan diet;
* Excessive alcohol consumption (on average >21 glasses/week for men and >14 glasses/week for women);
* Currently a research subject in another clinical trial;
* Having blood vessels that are too difficult for inserting a cannula/blood drawing'
* Having a hemoglobin level <8.5 mmol/l (men) or <7.5 mmol/l (women);
* Being a blood donor during the duration of the study;
* Not having a General Practitioner (GP);
* Being an employee of Wageningen University, division Human Nutrition and Health.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
postprandial glucose response (iAUC) per test product | 0-120 minutes
  iAUC glucose
small intestine microbiome | at baseline
  the relative composition (%) and the functional capacity (%) of the small intestine microbiota

SECONDARY OUTCOMES:
macronutrients in the small intestinal aspirates | 0-240 minutes
  amounts of carbohydrates, proteins, fats
presence and production of (bacterial) degradation products in the small intestinal aspirates | 0-240 minutes
  concentrations of organic acids and short-chain fatty acids
digestive enzymes in the small intestinal aspirates | 0-240 minutes
  concentrations of amylase
non-absorbable marker in the small intestinal aspirates | 0-240 minutes
  peg-4000 concentrations
blood HbA1c | 0-240 minutes
  concentrations of HbA1c
blood glucose | 0-240 minutes
  concentrations glucose (e.g. GLP-1, PYY)
blood insulin | 0-240 minutes
  concentrations of insulin
blood glucagon | 0-240 minutes
  concentrations of glucagon
blood total triglycerides | 0-240 minutes
  concentrations of triglycerides
blood total free fatty acids | 0-240 minutes
  concentrations of free fatty acids
plasma gut hormones | 0-240 minutes
  concentrations of gut hormones (e.g. GLP-1, PYY)
breath 13C-lactosyl ureide | 0-240 minutes
  concentrations of 13C-lactosyl ureide
breath hydrogen | 0-240 minutes
  concentrations of hydrogen (ppm)
breath methane | 0-240 minutes
  concentrations of methane (ppm)
Oral microbiome composition | baseline
  microbiota relative composition (%)
Salivary α-amylase | 0-240 minutes
  concentrations of a-amylase
Fecal microbiota composition | baseline
  microbiota relative composition (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No